CLINICAL TRIAL: NCT06126094
Title: Benefits of Alcoholic Hangover Medicine Myrkl
Brief Title: Benefits of Alcoholic Hangover Medicine
Acronym: BLAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Gut Microbiome Center (Centar za crijevni mikrobiom) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BLAM123
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Microbiome
Keywords: Microbiota; Probiotics; Alcohol; Cognitive behaviour
MeSH Terms: interventions — Dextrins

STUDY DESIGN:
Intervention Model Description: The test subjects receive capsules of probiotics and palcebo in marked bags and take one or the other arbitrarily without being told what is in which bag. Likewise, the researchers do not know whether the subjects took the probiotic or the placebo.
Who Masked: Participant, Investigator
Masking Description: The test subjects receive capsules of probiotics and palceb in marked bags and take one or the other arbitrarily without being told what is in which bag. Likewise, the researchers do not know whether the subjects took the probiotic or the placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Participants will consume 800 mg of probiotic Myrkl before consuming alcohol in the form of one capsule. (Myrkl, De Fair Medical, Stockholm, Sweden). This formulation contains AB001™, and one capsule (800mg) consists of:
  * 560 mg of naturally fermented rice bran
  * Bacillus subtilis
  * B. coagulans
  * L-cysteine
  * dextrin
  * 36 mg of excipients: magnesium stearate salts, calcium phosphate, potassium phosphate
  Interventions: Dietary Supplement: Myrkl
- Placebo (Experimental): The subject who consumed 800 mg of placebo- dextrin (maltodextrin) in the form of two capsules before consuming alcohol.
  Interventions: Dietary Supplement: dextrin

INTERVENTIONS:
Dietary Supplement: Myrkl — The subject of the test will be supplementation with precise probiotic for hangovers (Myrkl, De Fair) in the form of one pill of 800 mg
  Arms: Probiotic
Dietary Supplement: dextrin — The subject of the test will be supplementation with placebo (maltodextrin) in the form of two pills (each 400 mg)
  Arms: Placebo

SUMMARY:
Myrkl is advertised as a dietary supplement for use before alcohol consumption that is effective in prevention of side effects during the next day. With this research, the investigators want to determine the impact of the mentioned dietary supplement on the intestinal microbiome. For this purpose, the research was designed in three phases before, during and after the research as a double blind trial. In doing so, the subjects take a stool sample before and after the intervention and during the intervention, fill out questionnaires and undergo cognitive tests. At the same time, they give a blood sample after the intervention. After the results of the analysis are due, the researchers enter the data into the for that the predicted Access table (rel. representation of genera/genera/species, average results by questionnaires). The entered data is processed as part of statistical analysis.

DETAILED DESCRIPTION:
A "cure" for an alcoholic hangover has been put on the market, that is, it relieves the symptoms and ailments hangover alcohol (https://www.myrkl.com/). This medicine contains probiotic strains in its formulation (Bacillus subtilis, Bacillus coagulans). Myrkl has been advertised as a dietary supplement for use before alcohol consumption that is effective in prevention of side effects during the next day. The manufacturer claims that after taking Myrkl participants feel fresh even after a "long night". In addition to the probiotics mentioned above, Myrkl also contains L-cysteine and vitamins B12. The formula is said to be activated in the intestines. The manufacturer states that 77 of users are satisfied product and how it is completely natural. It is recommended to take two capsules two hours before consumption alcohol. With this research, the investigators wanted to determine the taxonomic changes within the intestinal microbiome after the intervention. In addition, the investigators wanted to determine changes in the subjective impression of a hangover measured by a validated questionnaires. The research was designed as a double-blind placebo-controlled intervention study twins (controlled for age, sex, cohabitation, genetics).

Before the start of the intervention, the test subjects will be instructed to eat the same diet during the 48 hours before beginning of each intervention. The subjects will keep a food diary for two days in order to accurately evaluated the nutritional status. The key is that both subjects consume the same food in both times before the intervention. The food intake itself is determined by the respondents independently.

After the intervention, the respondents will fill out a selection of questionnaires created in the form using the link a special online document (Project BLAM, Forms, Microsoft, USA) that will evaluate theirs alcoholic hangover. In order to evaluate the dynamics of the hangover, the test subject will again every 2 hours fill out the questionnaire (6 evaluations in total - waking up, 2, 4, 6, 8 and 10 hours after waking up). The result of each questionnaire is obtained by calculating the arithmetic mean of all answers (0-5, 0-10). Using all questionnaire was approved by the publisher and the English version will be used. Questionnaires were used https://forms.office.com/Pages/DesignPageV2.aspx subpage=design&FormId=hN0190t4UESOZ73jM ACw9LJ5ROlYHHVMuwYZ6ti3GaRUOEZEUVhSNDlPVjMwT1ZJVUFWTjQ3QldYRC4u&Token=fcda6871a b5d4009b779536b561d8dfb :

* Alcohol Hangover Questionnaire (AHQ)
* Alcohol Hangover Severity Scale (AHSS)

Materials The subject of the test will be supplementation with a precise probiotic for hangovers (Myrkl, De Fair

Medical, Stockholm, Sweden). This formulation contains AB001™, and one capsule (800mg) consists of:

* 560 mg of naturally fermented rice bran
* Bacillus subtilis
* B. coagulans
* L-cysteine
* dextrin
* 36 mg of excipients: magnesium stearate salts, calcium phosphate, potassium phosphate The CFU per strain in the formulation is minimal (ask the manufacturer). The probiotic comes in capsule form blister, stored at room temperature. An 800 mg capsule containing dextrin (maltodextrin) will be used for the placebo. It's a placebo dose also two capsules of 800 mg each.

The recommended intake will be two capsules exactly two hours before alcohol consumption. Control entry will be through a video diary.

Methods Analyzes of the intestinal microbiome Since the impact of probiotics on the intestinal microbiome will be measured before and after the investigated intervention two analyzes of the intestinal microbiome will be carried out on Day 0, i.e. on the day of the start of the intervention and Day 1, the day after the intervention. The BIOMES sampling kit will be used for the analysis, and intest.pro. The analysis will be performed on a sample of the first morning stool that the test subjects will take independently in home conditions Day 0 and Day 1. Samples will be delivered to the company's laboratory by logistics service BOMES (BIOMES GmbH, Wildau, Germany) where next-generation sequencing of 16s will be performed ribosomal RNA and bioinformatic analysis of the results (review of taxonomy and functionality). These results will be delivered to the researchers.

Statistical analysis Statistical data processing will analyze the changes in both test subjects, B1 and B2, taking taking into account whether the intervention was verum (V) or placebo (P). Upon maturity descriptive and inferential statistics will be made of the results using the appropriate program (Statistica, Palo Alto, USA). For normally distributed data, use the Kolmogorov-Smirnoff test will be the average and standard deviation, and for the second group the median and percentiles. To analyze the hypothesis treatment Mann-Whitney test and paired t-test will be used. Statistically significant will be considered p- values less than 0.05.

The research is divided into three phases - before the intervention, intervention, and after interventions. Alcohol is administered during the intervention. The respondents choose the drink they want consumed in two categories: welcome drink - žestice, brandy, liqueur, wormwood, evening drink - gemišt, wine, beer, gin and tonic, juice and juice.

Before intervention:

* the test subjects took the tests and research material at the Sky Office reception
* 48 hours before the intervention, they monitor their diet through a diary
* both test subjects eat absolutely identical food before each intervention
* on Day 0 they take the first stool sample (test A, test C), ideally the morning stool/the first stool
* do not consume any alcohol
* two hours before the planned intervention, say 6:30 p.m., that means around 4:30 p.m. they take a capsule with 1 dl water

Intervention:

* the subjects come to the recording on Day 0 around 18.00 in the CCM area, the conference room
* from 18.00 to 18.30 is preparation for recording
* at 6:30 p.m. the first sip of alcohol follows - a welcome drink (zestica, liqueur)
* around 6:40 p.m. the drinks of the evening follow (gemišt, gin and tonic, beer, wine)
* the first interview follows in terms of checking the degree of intoxication (cognitive tests 1-25/quiz)
* around 7:00 p.m., the first cut follows - a welcome drink
* around 7:10 p.m., another drink in the evening
* a second conversation follows in terms of checking the degree of intoxication (cognitive tests 1-25/quiz)
* during the second interview, the interviewees have the opportunity to eat something small (meal/sandwich)
* around 19.10 the last drink of the evening goes, possibly. and a welcome drink
* a third interview follows in terms of checking the degree of intoxication (cognitive tests 1-25/quiz)
* Human Lab takes a blood sample to determine blood ethanol, which CCM employees will take to HKA KBSD same evening immediately

After the intervention:

* after waking up and then within two hours, the subjects fill out the questionnaire: https://forms.office.com/Pages/ResponsePage.aspx?id=hN0190t4UESOZ73jMACw9LJ5ROlYH HVMuwYZ6ti3GaRUOEZEUVhSNDlPVjMwT1ZJVUFWTjQ3QldYRC4u
* the morning stool or the first stool after the intervention should be sampled on Day 1
* on Day 1 around 18.00 arrival for filming at the same place
* from 18.00 to 19.00 a conversation about how they feel and whether they think they received a placebo or a probiotic.

After the end of the cycle and the arrival of the results of the analysis, the researchers enter the data into the for that predicted Access table (rel. representation of genera/genera/species, average results by questionnaires). The entered data is processed as part of the statistical analysis in the previously explained manner. In these last steps student, research assistants may be involved.

ELIGIBILITY:
Inclusion Criteria:

• fraternal twins who live and work together

Exclusion Criteria:

* consumption of other probiotics, antibiotics 30 days before the research
* Inability to drink alcohol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Both participants should be female twins
Enrollment: 2 (Estimated)
Dates: Start 2023-10-31 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome composition | one month
  The impact of Myrkl on gut microbiome shall assessed through monitoring of relative taxonomic abundance of bacteria that compose gut microbiota from samples taken day before the intervention and after the intervention.
  The composition of the intestinal microbiota will be determined by sequencing the 16s rRNA bacteria in the stool sample. Subjects take a sample with a sterile cotton swab by wiping stool with toilet paper in their home on a given day research. The sample is stored in a tube with a buffer liquid so that the sample can be stored and transported at room temperature temperature. The test sample is transported by air to the laboratory of Biomes NGS Gesellschaft mit beschränkter Haftung, Wildau, Germany.

SECONDARY OUTCOMES:
the subjective impression of a hangover | one month
  In order to validate the subjective impression of a hangover, the subjects will fill out the Alcohol Hangover Questionnaire (AHQ) several times.

OTHER OUTCOMES:
other approach of impression of a hangover | one month
  n order to validate the subjective impression of a hangover, the respondants will fill out the Alcohol Hangover Severity Scale (AHSS) several times.

CONTACTS AND LOCATIONS:
Overall Officials: Andrija Karačić, dr.med, Study Director — Centar za crijevni mikrobiom
Locations (1):
- Gut Microbiome Center, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Chronic Uptake of A Probiotic Nutritional Supplement (AB001) Inhibits Absorption of Ethylalcohol in the Intestine Tract - Results from a Randomized Double-blind Crossover Study — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7141364/
- See also: Chronic Uptake of A Probiotic Nutritional Supplement (AB001) Inhibits Absorption of Ethylalcohol in the Intestine Tract - Results from a Randomized Double-blind Crossover Study — https://pubmed.ncbi.nlm.nih.gov/35769391/